CLINICAL TRIAL: NCT00352859
Title: A Randomized Discontinuation Trial to Determine the Clinical Benefit of Continuation of Sorafenib Following Disease Progression in Patients With Advanced Renal Cell Carcinoma
Brief Title: Phase IV Randomization to On-Going Treatment to Evaluate Sustained Sorafenib
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12178
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: Cancer; Renal Cell Cancer; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib; Interferons; Gemcitabine; Single Person

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006) with addition of gemcitabine or interferon
- Arm 2 (Experimental)
  Interventions: Drug: Gemcitabine or Interferon (only)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) with addition of gemcitabine or interferon — Continue sorafenib with addition of gemcitabine or interferon
  Arms: Arm 1
Drug: Gemcitabine or Interferon (only) — Discontinue Sorafenib and receive Gemcitabine or Interferon only
  Arms: Arm 2

SUMMARY:
The purpose of this study is to see if taking interferon or gemcitabine along with sorafenib will stop the advanced renal cell cancer from becoming worse in some people. To do this, sorafenib along with gemcitabine or interferon will be compared to treatment with gemcitabine or interferon alone. More safety information on sorafenib will be also collected. About 260 patients with progressed renal cell cancer will be in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients above 18 years of age with advanced RCC who have received sorafenib as their first and only systemic anti-tumor therapy for RCC prior to randomization
* Patients must have previously tolerated a minimum dose of sorafenib 400 mg daily for at least six weeks prior to study entry and have radiographically documented progressive disease while on sorafenib
* Patients must have experienced clinical benefit, partial response, complete response or stable disease during their previous course of sorafenib therapy
* Life expectancy > 12 weeks
* Patients must meet the Memorial Sloan-Kettering Cancer Center (MSKCC) risk category of low or medium at randomization
* Patients must give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Patients must have at least one uni-dimensional measurable lesion by CT-scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients must not have brain metastases
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* In addition, the following patients may be included, provided all other inclusion and exclusion criteria are met

  * Patients who have received the vaccines cG250 (monoclonal antibody to carbonic anhydrase IX) or HSPPC-96 (Heat Shock Protein Peptide Complex 96) are eligible provided that they have received no other systemic anti-cancer therapy
  * Patients who were enrolled in the ARCCS treatment protocol

Exclusion Criteria:

* Patients must not have experienced more than three weeks from documented disease progression to randomization
* Any medical condition requiring the use of systemic corticosteroids during IFN therapy
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated within the last three years prior to study entry
* Severe renal impairment or receiving dialysis
* More than a two week interruption in sorafenib dosing immediately prior to randomization
* Patients with a best response of disease progression on their previous course of sorafenib
* Patients who meet the MSKCC high risk category at randomization
* Hemorrhagic episode >= Grade 2 NCI CTC AE v3.0 within last six months
* History of cardiac disease: congestive heart failure> NYHA class 2; active cardiovascular disease (MI more than six months prior to study entry is allowed); cardiac arrhythmia requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
* Active clinically serious bacterial or fungal infections (>= Grade 2 NCI CTCAE v3.0)
* Known history of Human Immunodeficiency Virus (HIV) infection or chronic hepatitis B or C
* Symptomatic metastatic brain or meningeal tumors unless the patient is > six months from definitive therapy, has a negative CNS imaging study within four weeks of study entry, and is clinically stable off steroids. The patient must not be undergoing acute steroid taper
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* Ongoing substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial, including history of sensitivity to E. coli-derived products
* Any condition that is unstable or that could jeopardise the safety of the patient and his/her compliance in the study. Patients with a history of severe depression; patients with clinically significant active autoimmune disorders; history of organ allograft
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days of the start of study treatment. Both men and women enrolled in this trial must use adequate birth control measures during the course of the trial
* Patients who have had a significant surgical procedure within the past four weeks are excluded

Excluded Therapies and Medications, Previous and Concomitant:

* Any prior or concurrent systemic anti-cancer therapy including chemotherapy, monoclonal antibodies, hormonal therapy or investigational therapy, except for bisphosphonates and sorafenib
* Biological response modifiers, such as G-CSF or GM-CSF, within three weeks prior to study entry or during study. G-CSF and other hematopoietic growth factors may only be used in the management of acute toxicity such as febrile neutropenia when medically indicated or at the discretion of the Investigator. However, they may not be substituted for a required dose reduction of any study drug
* Patients taking erythropoietin are permitted provided no dose adjustment is undertaken within two months prior to the study or during the study
* Concomitant rifampicin or St. John's Wart
* Palliative therapy will be allowed, patients may receive palliative and supportive care for any underlying illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-08; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | After 192 progression or death events

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | After start of treatment
Overall Best Response | Until 30 days after termination of active therapy
Duration of response | Time from initial Response to documented Tumor Progression
Time to response | Time from the date of randomization to date that an objective tumor response (PR or CR) according to RECIST criteria is first documented
Overall Survival (OS) | Time from the date of randomization to date of death
Adverse Event Collection and Tolerability | Throughout the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kansas City, Missouri, United States